CLINICAL TRIAL: NCT02119936
Title: Feasibility of Heart Rate Variability Biofeedback as a Stress Reduction Tool for Hospitalized Pregnant Women at the University of North Carolina at Chapel Hill (UNC-CH)
Brief Title: Feasibility of Heart Rate Variability Biofeedback With In-patient Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-2051
Record Dates: First submitted 2014-04-16; First posted 2014-04-22 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-05

CONDITIONS: Maternal Stress; Maternal Anxiety; Maternal Health Services
Keywords: Stress; Anxiety; Mental Health; Mental Health Services; Maternal Mental Health
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heart Rate Variability Biofeedback Tool (Experimental): Intervention: Participants will be taught how to use the Heart Rate Variability Biofeedback tool (emWave 2) as a mechanism to reduce stress and anxiety, then use the tool, coupled with deep breathing exercises, to visualize their stress reduction.
  Interventions: Behavioral: Heart Rate Variability Biofeedback Tool

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback Tool — The Heart Rate Variability Biofeedback tool (emWave 2) will capture heart rate variability (HRV) before and after deep breathing exercises are used among participants. Participants will be able to visualize changes in their HRV and then fill-out self-reported anxiety measures to determine if the breathing exercises and visualization of HRV affected anxiety.
  Other Names: emWave 2 (Heartmath)

SUMMARY:
Purpose: The investigators plan a feasibility study on an easily disseminated biofeedback tool to reduce stress among hospitalized and expecting mothers. Converging evident suggests that Heart Rate Variability Biofeedback (HRVB) can improve the threshold of stress management and improve executive functioning. Additionally HRVB has been shown to significantly reduce anxiety features in women suffering from perinatal depression. The investigators hypothesize that HRVB will reduce stress levels among expecting mothers hospitalized for pregnancy complications, who are at high risk for depression and anxiety.

Participants: Expecting mothers hospitalized for pregnancy complication, who are at high risk for depression and anxiety.

Procedures: The investigators plain to use a heart rate variability biofeedback tool to measure stress reduction in hospitalized expectant mothers. This tool will be coupled with validated surveys and scales, high frequency heart rate variability, saliva samples, and qualitative interviews to quantify the reduction in stress from the HRVB tool.

DETAILED DESCRIPTION:
Background and Significance: Hospitalization during pregnancy is an unexpected interruption in the prenatal period that causes increased maternal anxiety and stress(MacMullen 1992). In a study of 129 women hospitalized for pregnancy complications, 25 met criteria for major depressive disorder(Brandon 2008). Such maternal depression is a risk factor for perinatal complications ranging from morbidity and mortality to neuropsychological developmental delays in the offspring(Poehlmann 2001). To date, however, few easily disseminated strategies have been identified to reduce stress among pregnant women.

To address this gap, the investigators plan a feasibility study of an easily-disseminated biofeedback tool to reduce stress among hospitalized expecting mothers(Beckham 2013). Converging evidence suggests that Heart Rate Variability Biofeedback (HRVB) can improve stress management and executive functioning (Association for Applied Psychophysiology and Biofeedback Inc 2011). Additionally, HRVB has recently been shown to reduce anxiety features in women suffering from perinatal depression at UNC (Beckham 2013). The investigators hypothesize that HRVB will reduce stress levels among expecting mothers hospitalized for pregnancy complications, who are at high risk for depression and anxiety(Brandon 2008).

Objectives:

1. To determine the feasibility of using HRVB among hospitalized pregnant women
2. To measure the association between use of HRVB and maternal state anxiety.
3. To measure the association between use of HRVB, biological markers of stress, indexed by salivary cortisol and oxytocin, and high frequency heart rate variability, measured using research-quality instruments
4. To measure the effectiveness of HRVB in women with varying levels of clinical depression and anxiety

Study Design & Methods: The investigators plan a pilot study to recruit 30 pregnant women who are receiving care on the antepartum floor of the North Carolina Women's Hospital.

At the baseline session,the investigators will consent each participant and then screen her for depression or anxiety. This screen will involve using the M.I.N.I Depression Module and the Edinburgh Postnatal Depression Screen (EPDS). Both assessments will be scored at baseline to determine if the participant has severe, moderate, or no clinical depression or anxiety. The investigators will also record if the participant is on anxiety or depression medication as apart of our screen. The investigators will also notes any medications given for other mental illness.

Once this screen is complete, the investigators will collect sociodemographic information and then proceed teach all the participants about biofeedback, how to use the HRVB device, coupled with deep breathing techniques to detach from stressful thoughts. The HRVB intervention will be administered by Carole Swanson, a registered nurse with extensive experience in maternity care, will complete the HeartMath® Interventions Certification Program(HeartMath LLC 2013). The certification provides detailed instruction on use of HRV Biofeedback for clinical care. The HeartMath device, the EmWave2, uses a heart rate sensor on the patient's earlobe to detect beat-to-beat variability, which is an index of vagal tone. The device is attached to a laptop computer to allow the user to view visual cues for deep breathing. The EmWave2 is currently used in clinical care in the inpatient psychiatry units at UNC hospitals.

Before and after each HRVB session, participants will complete three measures of current psychological distress (Spielberger State Anxiety Scale, Linear Analog Self Assessment, Warwick-Edinburgh Mental Well-Being scale). To measure biologic markers of stress, the investigators will collect saliva samples and measure blood pressure before and after administering HRVB. In addition information on the participants' high frequency heart rate variability will also be collected using the Single Channel 3991x Biolog, a research-quality measure of heart rate variability.

Participants will then be instructed to practice their deep breathing exercises for approximately ten minutes each day until the follow-up session and complete a brief log of these exercises. During this period participants will also be asked to complete validated inventories on perceived social support and life experiences (MOS Social Support Scale, Maternal Antenatal Attachment Scale and Adverse Childhood Experiences). At the follow up visit, approximately 5 to 7 days following the baseline session, administration of HRVB inventories on maternal mood, the saliva sample and measurement of high frequency heart rate variability will be repeated. The saliva sample will be used to measure salivary one or all of the following: oxytocin, alpha-amylase, and cortisol.

Finally the investigators will attempt a follow-up call with each participant six to eight weeks following discharge to measure continued use of HRVB techniques and satisfaction qualitative information on HRVB feasibility.

ELIGIBILITY:
Inclusion Criteria: Patients are eligible for the study if they fulfill all the inclusion criteria specified below:

1. Patient has signed the informed consent before any study specific procedures are performed.
2. Patient is a pregnant female over 18 years of age that is an in-patient on the UNC Women's Hospital antepartum floor.
3. Patient agrees to adhere to study requirements

Exclusion Criteria: Patients are not eligible for the study if they fulfill any of the exclusion criteria below:

1. Does not speak English.
2. Patient is not expected be on the antepartum floor of UNC Women's Hospital for at least 7 days.
3. Patient's healthcare provider does not want the patient to participate for medical safety purposes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Meltzer-Brody, MD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beckham AJ, Greene TB, Meltzer-Brody S. A pilot study of heart rate variability biofeedback therapy in the treatment of perinatal depression on a specialized perinatal psychiatry inpatient unit. Arch Womens Ment Health. 2013 Feb;16(1):59-65. doi: 10.1007/s00737-012-0318-7. Epub 2012 Nov 25. PMID 23179141
- [Result] Brandon AR, Trivedi MH, Hynan LS, Miltenberger PD, Labat DB, Rifkin JB, Stringer CA. Prenatal depression in women hospitalized for obstetric risk. J Clin Psychiatry. 2008 Apr;69(4):635-43. doi: 10.4088/jcp.v69n0417. PMID 18312059
- [Result] MacMullen N, Dulski LA, Pappalardo B. Antepartum vulnerability: stress, coping, and a patient support group. J Perinat Neonatal Nurs. 1992 Dec;6(3):15-25. doi: 10.1097/00005237-199212000-00004. No abstract available. PMID 1295961
- [Result] Poehlmann J, Fiese BH. The interaction of maternal and infant vulnerabilities on developing attachment relationships. Dev Psychopathol. 2001 Winter;13(1):1-11. doi: 10.1017/s0954579401001018. PMID 11346045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from the antepartum unit of the North Carolina Women's Hospital to participate in the study.
Groups:
- Heart Rate Variability Biofeedback: Intervention: Participants will be taught how to use the Heart Rate Variability Biofeedback (HRVB) tool (emWave 2) as a mechanism to reduce stress and anxiety, then use the tool, coupled with deep breathing exercises, to visualize their stress reduction.
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback
Started | 10
Completed | 0
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Population: 3 participants consented but delivered before baseline data was collected
Groups:
- Heart Rate Variability Biofeedback: Intervention: Participants will be taught how to use the Heart Rate Variability Biofeedback tool (emWave) as a mechanism to reduce stress and anxiety, then use the tool, coupled with deep breathing exercises, to visualize their stress reduction.
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Education status [Count of Participants; unit: Participants]
  Less than high school | 1
  High school diploma or GED equivalent | 2
  Some college credit, no degree | 4
  Associate's degree | 1
  Bachelor's degree | 1
  Graduate level degree | 1
Relationship status [Number; unit: participants] — More than one category could be selected so not representative of participant count
  participants
    Single/never married | 1
    Committed Relationship | 4
    Married | 4
    Divorced/separated | 2
    Widowed | 0
Insurance provider [Count of Participants; unit: Participants]
  Medicaid | 5
  Private Insurance | 5
  Tricare | 0
  Uninsured | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Using HRVB Among Hospitalized Pregnant Women
Description: The investigators will report rates of enrollment among women approached to join the study, rates of longitudinal data collection, and loss to follow-up.
Time Frame: Baseline, in-patient follow-up (5 to 7 days after baseline), and follow-up phone call (6 to 8 weeks post in-patient follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 10
Participants
  Participants enrolled | 10
  Participants with a 5-7 day inpatient follow-up | 0
  Participants with a follow up phone call | 0
  Participants completed | 0

2. Secondary Outcome: Change in State-Trait Anxiety Inventory From Baseline to In-patient Follow up (5-7 Days).
Description: State-trait anxiety scores range from 40-80 with higher scores indicative of greater anxiety
Time Frame: Baseline to in-patient follow-up (5 to 7 days in between)
Population: No in-patient follow up was completed due to patients moving off antepartum unit prior to meeting the 5-7 day in-patient criteria
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 0

3. Secondary Outcome: Association Between HRVB and High-Frequency Heart Rate Variability (HF-HRV)
Description: The investigators will measure HF-HRV in 1-minute segments during HRVB, and will test whether coherence score, as recorded by the HRVB device, correlates with HF-HRV.
Time Frame: Baseline to in-patient follow-up (5 to 7 days in between)
Population: HF-HRV data was not collected
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation of HRVB Feedback With Varying Levels of Clinical Depression and Anxiety
Description: The investigators will stratify our population based on the depression screen used at the baseline visit. These groups will include those with severe, moderate, or lack of depression. The investigators will then compare these groups to the finds from the surveys on maternal mood and the difference noticed among the groups due to the HRVB tools.
Time Frame: Baseline to in-patient follow-up (5 to 7 days in between)
Population: All participants were discharged from the antepartum unit prior to 5-7 days in-patient so these data were not collected.
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Linear Analog Self-Assessment (LASA) From Baseline to In-patient Follow up (5-7 Days).
Description: The Linear Analog Self-Assessment (LASA) form measures patient quality-of-life. Scores range from 6-30 with higher scores indicative of greater well-being.
Time Frame: Baseline to in-patient follow-up (5 to 7 days in between)
Population: All participants were discharged from antepartum unit prior to 5-7 days in-patient so these study data were not collected.
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Warwick Edinburgh Mental Well Being Scale From Baseline to In-patient Follow up (5-7 Days).
Description: The Warwick Edinburgh Mental Well Being Scale is a 14 item self-report measure assessing subjective well-being (1-5 scale). Higher values represent more positive mental well being. The summary measure is a sum of the 14 questions (not a mean). Summary values therefore range from 14-70.
Time Frame: Baseline to in-patient follow-up (5 to 7 days in between)
Population: All participants were discharged from the antepartum unit prior to 5-7 days in-patient so these study data were not collected.
Arm/Group | Heart Rate Variability Biofeedback
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No difference from clinicaltrials.gov definition
Arm/Group | Heart Rate Variability Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes